CLINICAL TRIAL: NCT00813501
Title: Evaluation of Clinical Utility of the Cylex ImmunKnow Assay in Hematopoietic Cell Transplantation
Brief Title: Immunologic Diagnostic Blood Test in Predicting Side-Effects in Patients Undergoing a Donor Stem Cell Transplant for Hematologic Cancer or Other Diseases
Status: Terminated | Type: Observational
Why Stopped: Terminated at the request of the study sponsor
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: David Senitzer, City of Hope Comprehensive Cancer Center
Other Study IDs: 07200; P30CA033572 (NIH); CHNMC-07200; CDR0000628793 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-12-20; First posted 2008-12-23 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Infection; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Therapy-related Toxicity
Keywords: graft versus host disease; infection; therapy-related toxicity; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Infections; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Hairy Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic | interventions — Immunosuppression Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: immunosuppressive therapy
Other: immunological diagnostic method
Procedure: allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Studying a diagnostic biomarker test in blood samples from patients who have undergone a donor stem cell transplant for cancer may help doctors plan treatment.

PURPOSE: This clinical trial is studying an immunologic diagnostic blood test to see how well it works in predicting side-effects in patients with hematologic cancer or other disorders who have undergone a donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the ability of the ImmuKnow® test to predict the onset and severity of acute or chronic graft-versus-host disease and/or measure the clinical effects of treatment.
* To evaluate the ability of the ImmuKnow test to predict the clinical response to immunosuppressive therapy.
* To evaluate the ability of the ImmuKnow test to predict infections among patients.

OUTLINE: Beginning on day 14 after allogeneic hematopoietic stem cell transplantation (HSCT), patients undergo blood sample collection at least once weekly for the first 100 days and then once to twice monthly for up to 1 year, in the absence of graft-versus-host disease (GVHD). If chronic or acute GVHD develops after day 100, more frequent blood sampling may occur. Blood sample collection is coordinated with the time of regular clinic visits to allow for evaluation of the clinical events recorded 2 weeks before and after the blood draw date. Blood samples are analyzed by the Cylex® and ImmuKnow® assays to measure global T-cell immune function and responsiveness to alterations in immunosuppressive post-HSCT therapy. Assay data obtained during the first 3 weeks and other post-transplant periods will be evaluated for possible correlations with clinical endpoints (i.e., GVHD incidence, rate of infection, and response to immunosuppressive therapy) to assess the predictive value of the assay.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematologic cancer or other disease
* Undergoing allogeneic hematopoietic stem cell transplantation

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing allogeneic hematopoietic stem cell transplantation at the City of Hope Medical Center
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Acute graft-versus-host disease (GVHD)
Grade of acute GVHD
Response criteria for treatment of acute GVHD
Chronic GVHD
Grade of chronic GVHD
Response criteria for treatment of chronic GVHD
Infections (i.e., bacterial, fungal, or viral)

CONTACTS AND LOCATIONS:
Overall Officials: David Senitzer, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States